CLINICAL TRIAL: NCT04916795
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, SINGLE DOSE STUDY TO INVESTIGATE THE PHARMACOKINETICS, PHARMACODYNAMICS, SAFETY AND TOLERABILITY OF VUPANORSEN ADMINISTERED SUBCUTANEOUSLY TO HEALTHY CHINESE ADULTS
Brief Title: A Study To Investigate The Pharmacokinetics, Pharmacodynamics, Safety And Tolerability Of Single Dose Vupanorsen In Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4491004
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — vupanorsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vupanorsen 80 milligram (mg) (Experimental): Participants will receive one, 0.8 milliliter (mL) subcutaneous injection with vupanorsen 100 mg/mL solution
  Interventions: Drug: Vupanorsen
- Vupanorsen 160 milligram (mg) (Experimental): Participants will receive two, 0.8 mL subcutaneous injections with vupanorsen 100 mg/mL solution
  Interventions: Drug: Vupanorsen

INTERVENTIONS:
Drug: Vupanorsen — 80 mg subcutaneous injection
  Arms: Vupanorsen 80 milligram (mg)
Drug: Vupanorsen — 80 mg subcutaneous injection
  Arms: Vupanorsen 160 milligram (mg)

SUMMARY:
This is a Phase 1, randomized, parallel-cohort, open-label study to characterize the pharmacokinetics, pharmacodynamics, safety and tolerability of vupanorsen following 80 mg and 160 mg single subcutaneous dose in healthy Chinese adults with elevated fasting triglyceride.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Chinese participants must be 18 to 65 years of age, inclusive, at the time of signing the ICD.

   * Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.
   * Chinese participant is defined as individuals currently residing in mainland China who were born in China and have both parents of Chinese descent.
2. Male and female Chinese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests (except for TG levels), and 12-lead ECG monitoring.
3. Fasting TG ≥ 90 mg/dL at Screening (up to 1 repeat allowed for TG and the second TG value will be used for the eligibility).
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
5. BMI of 17.5 to 35.0 kg/m2; and a total body weight >50 kg (110 lb).
6. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of human immunodeficiency virus (HIV) infection, syphilis, hepatitis B, or hepatitis C; positive testing for HIV, syphilis, HBsAg, or HCVAb. Prior Hepatitis B vaccination is allowed.
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
5. Previous administration with an investigational drug within 4 months or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
6. A positive urine drug test.
7. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * AST or ALT level ≥1.25 × ULN;
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
11. Blood donation (excluding plasma donations) of approximately 400 mL or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin-induced thrombocytopenia.
13. History of substance abuse within 12 months of the screening visit.
14. Pregnant females; breastfeeding females.
15. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
16. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wu X, Yu J, Ge B, Wang J, Han X, Zhang C, Mao X, Kalluru H, Bramson C, Terra SG, Liu J. A Randomized, Open-Label, Phase I, Single-Dose Study of Antisense Oligonucleotide, Vupanorsen, in Chinese Adults with Elevated Triglycerides. Drugs R D. 2024 Jun;24(2):253-262. doi: 10.1007/s40268-024-00467-5. Epub 2024 Jul 1. PMID 38949758
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4491004

RESULTS

PARTICIPANT FLOW:
Groups:
- Vupanorsen 80 mg: Participants were selected and categorized into the Vupanorsen 80 mg group and received a single 80 mg subcutaneous dose of vupanorsen on Day 1, followed by an on-site post-treatment evaluation on Days 8, 15, 30, 60 and 90.
- Vupanorsen 160 mg: Participants were selected and categorized into the Vupanorsen 160 mg group and received a single 160 mg subcutaneous dose of vupanorsen on Day 1, followed by an on-site post-treatment evaluation on Days 8, 15, 30, 60 and 90.
Period: Overall Study
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants enrolled and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.44 (7.13) | 36.22 (8.45) | 33.83 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time 0 to 24 Hours Post-dose (AUC24h) for Vupanorsen
Description: AUC24h is the area under the concentration-time profile from time 0 to 24 hour post-dose
Time Frame: 0 hour (predose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on day 1
Population: The analysis population refers to all participants enrolled and treated who had at least 1 of the vupanorsen pharmacokinetic (PK) parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(mcg*hr/mL)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
microgram*hour per milliliter(mcg*hr/mL) | 3.649 (35) | 10.82 (42)

2. Primary Outcome: AUC From Time 0 to 48 Hours Post-dose (AUC48h) for Vupanorsen
Description: AUC48h is the area under the plasma concentration-time profile from time zero to the quantifiable concentration 48 hours post-dose
Time Frame: 0 hour (predose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post dose
Population: The analysis population refers to all participants enrolled and treated who had at least 1 of the vupanorsen PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
mcg*hr/mL | 3.699 (34) | 10.91 (42)

3. Primary Outcome: AUC From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) for Vupanorsen
Description: AUClast is the area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast)
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
mcg*hr/mL | 3.950 (34) | 11.76 (39)

4. Primary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum plasma concentration observed from data
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
microgram per milliliter (μg/mL) | 0.5879 (62) | 1.810 (63)

5. Primary Outcome: AUC From Time 0 Extrapolated to Infinite Time (AUCinf) for Vupanorsen
Description: AUCinf is area under the plasma concentration-time profile from time zero extrapolated to infinite time
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 8 | 9
mcg*hr/mL | 4.081 (36) | 11.91 (39)

6. Primary Outcome: Time for Cmax (Tmax) for Vupanorsen
Description: Time for Cmax (Tmax) for vupanorsen
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
hour (hr) | 2.00 [1.50 to 3.00] | 2.00 [1.50 to 3.00]

7. Primary Outcome: Terminal Elimination Half Life (t½) for Vupanorsen
Description: terminal elimination half life (t½) for vupanorsen
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour (hr)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 8 | 9
hour (hr) | 475.9 (205.50) | 465.2 (131.50)

8. Primary Outcome: Apparent Clearance (CL/F) for Vupanorsen
Description: Apparent clearance for vupanorsen
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 8 | 9
liter per hour (L/hr) | 19.60 (36) | 13.43 (39)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F) for Vupanorsen
Description: Apparent volume of distribution for vupanorsen
Time Frame: 0 hour (predose), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose, and on days 8, 15, 30, 60 and 90
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 8 | 9
liter (L) | 12500 (37) | 8681 (48)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product or medical device, without regard to causality. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. AEs included SAEs and non-serious AEs. Treatment-related TEAEs were any untoward medical occurrence attributed to study treatment. Causality to study treatment was determined by the investigator.
Time Frame: Baseline through day 90
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
Participants
  All-causality | 3 | 5
  Treatment-related | 2 | 1

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Protocol-required safety laboratory assessments included chemistry, hematology, and urinalysis (and microscopy, if needed). Each parameter was evaluated against commonly used and widely accepted criteria.
Time Frame: Baseline through day 90
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
Participants | 5 | 5

12. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Values
Description: Vital sign data included blood pressure and pulse rate. Clinical significance was assessed by the investigator.
Time Frame: Baseline through day 90
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
Participants | 1 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Values
Description: Clinical significance of ECG data was assessed by the investigator.
Time Frame: Baseline through day 90
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

14. Secondary Outcome: Percent Changes From Baseline in Angiopoietin-Like 3 (ANGPTL3)
Description: Percent changes from baseline in ANGPTL3 on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the pharmacodynamic (PD) parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -13.88 (18.644) | -22.14 (15.103)
  DAY3 | -32.65 (22.375) | -43.56 (15.151)
  DAY8 | -59.65 (18.727) | -69.11 (13.462)
  DAY15 | -54.07 (21.893) | -69.48 (11.659)
  DAY30 | -48.66 (21.921) | -62.81 (18.873)
  DAY60 | -38.54 (23.440) | -53.33 (11.830)
  DAY90 | -12.69 (20.238) | -29.72 (15.587)

15. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Percentage changes from baseline in total cholesterol on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -1.50 (5.839) | -2.04 (6.238)
  DAY3 | -1.71 (9.012) | -0.71 (7.665)
  DAY8 | -18.89 (6.814) | -20.39 (8.526)
  DAY15 | -19.57 (12.554) | -21.85 (11.371)
  DAY30 | -10.46 (14.303) | -11.11 (7.976)
  DAY60 | -8.26 (16.712) | -1.76 (10.038)
  DAY90 | -5.10 (14.122) | -3.06 (7.317)

16. Secondary Outcome: Percent Changs From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Percentage changes from baseline in HDL-C on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -0.55 (3.636) | -0.79 (8.504)
  DAY3 | -3.81 (2.908) | -0.14 (9.771)
  DAY8 | -3.97 (13.335) | -9.16 (16.834)
  DAY15 | -3.33 (20.205) | -10.08 (16.485)
  DAY30 | 8.96 (18.824) | 3.70 (15.475)
  DAY60 | 8.19 (13.457) | 5.18 (15.265)
  DAY90 | 6.74 (14.464) | 5.92 (12.033)

17. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Percentage changes from baseline in LDL-C on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | 2.94 (9.247) | -0.63 (7.817)
  DAY3 | 1.91 (12.944) | 2.80 (11.548)
  DAY8 | -14.65 (9.005) | -12.10 (15.647)
  DAY15 | -14.95 (19.076) | -15.93 (16.486)
  DAY30 | -9.86 (22.385) | -6.03 (16.710)
  DAY60 | -12.77 (23.668) | 0.19 (15.380)
  DAY90 | -7.42 (19.649) | 2.97 (10.818)

18. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C)
Description: Percentage changes from baseline in VLDL-C on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -15.93 (18.320) | -1.16 (28.947)
  DAY3 | 5.68 (35.419) | -4.79 (45.277)
  DAY8 | -65.66 (19.581) | -72.26 (21.036)
  DAY15 | -62.44 (27.207) | -64.24 (31.482)
  DAY30 | -27.64 (40.099) | -53.51 (27.018)
  DAY60 | 11.09 (50.942) | 8.28 (77.143)
  DAY90 | -22.63 (58.405) | -51.39 (37.174)

19. Secondary Outcome: Percent Change From Baseline in Triglyceride
Description: Percentage changes from baseline in triglyceride on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -9.72 (15.235) | -5.86 (12.887)
  DAY3 | -10.03 (16.856) | -7.24 (26.804)
  DAY8 | -32.61 (16.422) | -52.47 (18.150)
  DAY15 | -41.91 (19.992) | -48.19 (16.491)
  DAY30 | -28.54 (20.289) | -44.14 (19.466)
  DAY60 | -19.55 (29.981) | -30.60 (23.585)
  DAY90 | 7.26 (59.830) | -21.26 (28.335)

20. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percentage changes from baseline in non-HDL on Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Time Frame: Day 1, Day 2, Day 3, Day 8, Day 15, Day 30, Day 60 and Day 90
Population: All participants enrolled and treated who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: percent change (%)
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 9 | 9
percent change (%)
  DAY2 | -1.39 (7.609) | -2.40 (6.649)
  DAY3 | -0.12 (12.865) | -0.89 (9.120)
  DAY8 | -22.58 (8.362) | -23.41 (8.368)
  DAY15 | -23.18 (15.173) | -25.37 (11.202)
  DAY30 | -15.33 (16.925) | -15.58 (10.089)
  DAY60 | -11.58 (22.194) | -3.89 (9.669)
  DAY90 | -8.32 (16.806) | -6.35 (7.602)

21. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (ApoA-I)
Description: Percentage changes from baseline in ApoA-I on Day 15, Day 60, and Day 90. This endpoint was terminated due to changes of development plan.
Time Frame: Day 1, Day 15, Day 60, and Day 90
Population: Study endpoint of percent changes from baseline in apolipoprotein A-1 (ApoA-I),apolipoprotein B (ApoB) total (including ApoB-48, ApoB-100), and apolipoprotein C-III (ApoC-III) on Day 15, Day 60, and Day 90, were terminated due to changes of development plan. No data were collected for these terminated endpoints.
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) Total (Including ApoB-48, ApoB-100)
Description: Percentage changes from baseline in ApoB total (including ApoB-48, ApoB-100) on Day 15, Day 60, and Day 90. This endpoint was terminated due to changes of development plan.
Time Frame: Day 1, Day 15, Day 60, and Day 90
Population: as for outcome 21
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-III (ApoC-III)
Description: Percentage changes from baseline in apolipoprotein C-III (ApoC-III) on Day 15, Day 60, and Day 90. This endpoint was terminated due to changes of development plan.
Time Frame: Day 1, Day 15, Day 60, and Day 90
Population: as for outcome 21
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through day 90
Arm/Group | Vupanorsen 80 mg | Vupanorsen 160 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vupanorsen 80 mg (N=9) | Vupanorsen 160 mg (N=9)
Palpitations (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04916795/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT04916795/SAP_001.pdf